CLINICAL TRIAL: NCT01153958
Title: The Use of Colposeptine in Bacterial Vaginosis. A Randomized, Controlled Study
Brief Title: Colposeptine for the Treatment of Bacterial Vaginosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200059-504
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Vaginosis, Bacterial
Keywords: Vaginosis, Bacterial; Colposeptine; Metronidazole
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colposeptine (A) (Experimental)
  Interventions: Drug: Colposeptine
- Metronidazole (B) (Active Comparator)
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Colposeptine — Colposeptine will be administered transvaginally at a dose of 1 capsule every day for 12 consecutive days
  Other Names: Chlorquinaldol-Promestriene Vaginal Capsules
  Arms: Colposeptine (A)
Drug: Metronidazole — Metronidazole will be administered orally at a dose of 400 mg twice a day for 7 days
  Arms: Metronidazole (B)

SUMMARY:
This is a prospective, randomized, controlled and multi-center trial to assess the use of colposeptine in female subjects with bacterial vaginosis. A total of 480 subjects were planned to be enrolled in various centers in China.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects in reproductive age and older than 18 year
* Subjects with normal sexual activity
* Subjects with symptoms such as vulva-vaginal irritation or abnormal vaginal discharge
* Subjects with Nugent Score greater than or equal to 7
* Subjects who are willing to use contraception
* Subjects who are willing to refrain from the use of other vaginal products throughout the study
* Subjects who sign informed consent form and agree to follow-up on time

Exclusion Criteria:

* Subjects without sexual activity
* Pregnant or lactating female subjects
* Subjects with a history of recurrent bacterial vaginosis
* Subjects diagnosed with trichomonas vaginitis，vulvovaginal candidiasis，chlamydia or gonococcus infection.
* Subjects who are unwilling to refrain from the ingestion of any alcoholic beverages during the 7 day course of oral metronidazole therapy
* Subjects who are under treatment by lithium, phenobarbitone, coumadine anticoagulant, cyclosporine or disulfiram by the time of inclusion (interactions with other products and metronidazole)
* Subjects who are undergoing systemic or topical treatment with antibiotics, steroids, immunosuppressive, cytostatic or antimetabolic agents by the time of inclusion
* Female subjects with a history of peripheral neuropathy
* Female subjects who have participated in another clinical trial or have taken an experimental drug within the past 30 days
* Subjects who are unable to give written informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Merck Serono Co., Ltd., China
Locations (5):
- China (5):
  - Peking University People's Hospital, Beijing
  - Second Hospital of West China Medical School, Sichuan University, Chengdu
  - Obstetrics & Gynaecology Hospital of Fudan University, Shanghai
  - Peking University Shenzhen Hospital, Shenzhen
  - Wuhan Union Hospital of China, Wuhan

RESULTS

PARTICIPANT FLOW:
Groups:
- Colposeptine: Colposeptine 1 capsule transvaginally daily for 12 consecutive days.
- Metronidazole: Metronidazole 400 milligram (mg) orally twice daily for 7 consecutive days
Period: Overall Study
Arm/Group | Colposeptine | Metronidazole
Started | 66 | 67
Completed | 30 | 35
Not Completed | 36 | 32
Not completed — Study Terminated | 36 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colposeptine | Metronidazole | Total
Number analyzed (Participants) | 66 | 67 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.11 (8.78) | 30.72 (7.06) | 31.41 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 67 | 133
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapse 2 Months Post-treatment
Description: Relapse: recurrence of the symptoms of bacterial vaginosis [BV] (Nugent score greater than or equal to 7, symptoms of vaginal irritation for example, pain, burning, odour or abnormal vaginal discharge) after a period of improvement. Nugent score was calculated by assessing for presence of large Gram-positive rods (Lactobacillus morphotypes; decrease in Lactobacillus scored as 0-4), small Gram-variable rods (Gardnerella vaginalis morphotypes; scored as 0-4), and curved Gram-variable rods (Mobiluncus species morphotypes; scored as 0-2). Total score range: 0-10. Score of 7-10 indicated BV.
Time Frame: 2 months post-treatment
Population: Full analysis set (FAS) population included all enrolled participants who used investigational product. 'N' (number of participants analyzed) signifies those participants who were evaluated for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Colposeptine | Metronidazole
Number analyzed (Participants) | 30 | 35
percentage of participants | 23.3 | 17.2

2. Secondary Outcome: Percentage of Participants With Relapse 1 Month Post-treatment
Description: as for outcome 1
Time Frame: 1 month post-treatment
Population: FAS population included all enrolled participants who used investigational product. 'N' (number of participants analyzed) signifies those participants who were evaluated for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Colposeptine | Metronidazole
Number analyzed (Participants) | 25 | 28
percentage of participants | 16.0 | 10.7

3. Secondary Outcome: Change From Baseline in Nugent Score at 2 Months Post-treatment
Description: Nugent score was calculated by assessing for presence of large Gram-positive rods (Lactobacillus morphotypes; decrease in Lactobacillus scored as 0-4), small Gram-variable rods (Gardnerella vaginalis morphotypes; scored as 0-4), and curved Gram-variable rods (Mobiluncus species morphotypes; scored as 0-2). Total score range: 0-10. Score of 7-10 indicate bacterial vaginosis.
Time Frame: Baseline and Month 2 post-treatment
Population: FAS population included all enrolled participants who used investigational product. 'n' signifies those participants who were evaluated for this measure at the time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colposeptine | Metronidazole
Number analyzed (Participants) | 66 | 67
units on a scale
  Baseline (n= 66, 67) | 7.86 (0.58) | 8.01 (0.59)
  Change at Month 2 (n= 25, 29) | 3.20 (2.12) | 4.03 (2.71)

4. Secondary Outcome: Change From Baseline in Number of Participants With Each Grade of Lactobacilli at 2 Months Post-treatment
Description: The grades of Lactobacilli in vaginal discharge were Grade 1 (Normal): Lactobacillus morphotypes predominate; Grade 2 (Intermediate): Mixed flora with some Lactobacilli present, but Gardnerella or Mobiluncus morphotypes also present; Grade 3 (Bacterial Vaginosis): Predominantly Gardnerella and/or Mobiluncus morphotypes, few or absent Lactobacilli.
Time Frame: Baseline and Month 2 post-treatment
Population: FAS population included all enrolled participants who used investigational product. 'N' (number of participants analyzed) signifies those participants who were evaluated for this measure. 'n' signifies those participants who were evaluated for this measure at the time point.
Measure: Number; unit: participants
Arm/Group | Colposeptine | Metronidazole
Number analyzed (Participants) | 66 | 66
participants
  Baseline, Grade 1 (n= 66, 66) | 0 | 0
  Baseline, Grade 2 (n= 66, 66) | 3 | 1
  Baseline, Grade 3 (n= 66, 66) | 63 | 65
  Month 2, Grade 1 (n= 25, 29) | 11 | 9
  Month 2, Grade 2 (n= 25, 29) | 7 | 14
  Month 2, Grade 3 (n= 25, 29) | 7 | 6

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Time Frame: Up to 2 months post-treatment
Population: Safety population included all randomized participants who used the investigational product at least once.
Measure: Number; unit: participants
Arm/Group | Colposeptine | Metronidazole
Number analyzed (Participants) | 66 | 67
participants | 8 | 8

6. Secondary Outcome: Percentage of Participants Cured
Description: Cure was defined as Nugent score less than 7, no symptoms of vaginal irritation (for example, pain, burning, odour or abnormal vaginal discharge). Nugent score was calculated by assessing for presence of large Gram-positive rods (Lactobacillus morphotypes; decrease in Lactobacillus scored as 0-4), small Gram-variable rods (Gardnerella vaginalis morphotypes; scored as 0-4), and curved Gram-variable rods (Mobiluncus species morphotypes; scored as 0-2). Total score range: 0-10. Score of 7-10 indicated bacterial vaginosis.
Time Frame: 1 week post-treatment
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Colposeptine | Metronidazole
Number analyzed (Participants) | 48 | 45
percentage of participants | 22.9 | 17.8

ADVERSE EVENTS:
Time Frame: Baseline up to 2 months post-treatment
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Colposeptine | Metronidazole
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/67
Other Adverse Events (participants affected / at risk) | 8/66 | 10/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colposeptine (N=66) | Metronidazole (N=67)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Vulvovaginal Candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Endodontic Procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Vulvovaginitis Trichomonal (Infections and infestations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (2) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other